CLINICAL TRIAL: NCT04429789
Title: Waking Hypnosis in the Treatment of MS-related Fatigue: Pilot and Feasibility Study
Brief Title: Waking Hypnosis in the Treatment of MS-related Fatigue
Acronym: POWER-UP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, M. Elena Mendoza, Principal Investigator, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00007428; PP-1904-33857 (Other Grant/Funding Number: National Multiple Sclerosis Society)
Record Dates: First submitted 2020-05-11; First posted 2020-06-12 (Actual); Last update posted 2021-05-03 (Actual); Status verified 2021-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: Single-center, single-blind three-group randomized (1:1:1) controlled trial (RCT) comparing two hypnosis interventions to waitlist control efficacy for MS-related fatigue.
Who Masked: Outcomes Assessor
Masking Description: Research assistant administering the telephone assessments is blinded to participant treatment intervention while the clinician conducting the treatment sessions is blinded to participant responses provided during telephone assessments. The only instance where we may unblind staff members to assessment or treatment data (depending on what the staff member is responsible for) will be at the end of the study, after data collection has been completed. At that point, the staff member conducting telephone assessments may be allowed to know which interventions participants were assigned to, and the clinician conducting treatment sessions may be allowed to access assessment data if a staff member were to assist in data cleaning or data analysis. Participants are blind to study hypotheses and will not be told which intervention is expected to yield what results. Participants may be unblinded if/when we disseminate findings (e.g., in a published manuscript) related to this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active-Alert Hypnosis (Experimental)
  Interventions: Behavioral: Active-Alert Hypnosis
- Traditional Hypnosis (Experimental)
  Interventions: Behavioral: Traditional Hypnosis
- Wait-List Control (No Intervention): Participants in this arm will continue their usual care for fatigue. The therapist will notify participants assigned to Usual Care via the participant's preferred mode of communication (phone, U.S. mail, or email). People assigned to usual care will be encouraged to continue using the health care services available to them to address their fatigue. The study therapist will emphasize the importance of completing the outcome assessments. Following the completion of their final assessment (3 month follow-up); these individuals will be offered their choice of the two hypnosis treatments.

INTERVENTIONS:
Behavioral: Active-Alert Hypnosis — Participants in this arm will receive four one-hour weekly sessions that will include training in a rapid self-hypnosis method. Participants will learn how to use waking hypnosis to manage fatigue using exercises with sensory experiences.
  Arms: Active-Alert Hypnosis
Behavioral: Traditional Hypnosis — Participants in this arm will receive four one-hour weekly sessions where participants will learn how to use hypnosis along with relaxation. The exercises and suggestions included in the training will be adapted from the protocol used in a series of studies on the efficacy of self-hypnosis training for the management of chronic pain in persons with disabilities, and from a therapist guide of procedures and hypnotic suggestions for chronic pain.
  Arms: Traditional Hypnosis

SUMMARY:
The proposed study is a single-center, single-blind three-group randomized (1:1:1) controlled trial (RCT) comparing two hypnosis interventions to waitlist control efficacy for MS-related fatigue.

DETAILED DESCRIPTION:
This project will test the efficacy of two different hypnosis approaches for improving MS-related fatigue that have shown to be beneficial for individuals with cancer and other medical conditions in the management of their symptoms. One of these methods, the active-alert hypnosis has helped people to manage fatigue and may have important advantages over the more traditional relaxation hypnotic approaches in the treatment of fatigue, since the hypnotic inductions and the self-hypnosis methods use activation instead of relaxation. Therefore, the goals of this study are to determine if a comparison study of these two hypnotic conditions is feasible, and, if so, to determine which treatment may be more effective for helping individuals with MS gain more control over fatigue. Additionally, it will explore the mechanisms of these two approaches to hypnosis treatment to determine which might be most helpful to individuals with MS and fatigue.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MS;
* Adults 18 years of age or older;
* Bothersome fatigue (defined as the presence of chronic, problematic fatigue that, in the opinion of the patient, has interfered with their daily activities for ≥ 3 months and average Fatigue Severity Scale score > to 4 at screening);
* Ability to read, speak, and understand English and/or Spanish.

Exclusion Criteria:

* Exclusion criteria will be evidence for significant psychopathology that would interfere with study participation, including current suicidal ideation with intent, active psychosis or hallucinations, or severe cognitive impairment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-05-27 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Fatigue Self Efficacy | Assessed via telephone within a 1-week period at baseline (prior to randomization)
  Multiple Sclerosis-Fatigue Self-Efficacy scale
Fatigue Self Efficacy | Third week: mid-treatment (after second session)
  Multiple Sclerosis-Fatigue Self-Efficacy scale
Fatigue Self Efficacy | Fifth week: post-treatment (after fourth session)
  Multiple Sclerosis-Fatigue Self-Efficacy scale
Fatigue Self Efficacy | 4 months: 3 month follow-up
  Multiple Sclerosis-Fatigue Self-Efficacy scale
Fatigue Severity | Assessed via telephone within a 1-week period at baseline (prior to randomization)
  Fatigue Severity Scale (FSS) score
Fatigue Severity | Third week: mid-treatment (after second session)
  Fatigue Severity Scale (FSS) score
Fatigue Severity | Fifth week: post-treatment (after fourth session)
  Fatigue Severity Scale (FSS) score
Fatigue Severity | 4 months: 3 month follow-up
  Fatigue Severity Scale (FSS) score

SECONDARY OUTCOMES:
Psychological and Physical Function | Assessed via telephone within a 1-week period at baseline (prior to randomization)
  PROMIS Physical Function SF score
Psychological and Physical Function | Third week: mid-treatment (after second session)
  PROMIS Physical Function SF score
Psychological and Physical Function | Fifth week: post-treatment (after fourth session)
  PROMIS Physical Function SF score
Psychological and Physical Function | 4 months: 3 month follow-up
  PROMIS Physical Function SF score
Activity Level | Assessed via telephone within a 1-week period at baseline (prior to randomization)
  IPAQ: International Physical Activity Questionnaire SF score
Activity Level | Third week: mid-treatment (after second session)
  IPAQ: International Physical Activity Questionnaire SF score
Activity Level | Fifth week: post-treatment (after fourth session)
  IPAQ: International Physical Activity Questionnaire SF score
Activity Level | 4 months: 3 month follow-up
  IPAQ: International Physical Activity Questionnaire SF score
Suggestibility | Within a 1-week period at baseline (prior to randomization)
  Barber Suggestibility Scale score
Suggestibility | Fifth week: post-treatment (after fourth session)
  Barber Suggestibility Scale score
Attitudes towards hypnosis | Assessed via telephone within a 1-week period at baseline (prior to randomization)
  Valencia Scale of Attitudes and Beliefs toward Hypnosis -Client version
Attitudes towards hypnosis | Third week: mid-treatment (after second session)
  Valencia Scale of Attitudes and Beliefs toward Hypnosis -Client version
Attitudes towards hypnosis | Fifth week: post-treatment (after fourth session)
  Valencia Scale of Attitudes and Beliefs toward Hypnosis -Client version
Attitudes towards hypnosis | 4 months: 3 month follow-up
  Valencia Scale of Attitudes and Beliefs toward Hypnosis -Client version
Treatment Outcome Expectancy | Assessed via telephone within a 1-week period at baseline (prior to randomization)
  Treatment Expectancy Scale
Sleep Quality | Assessed via telephone within a 1-week period at baseline (prior to randomization)
  PROMIS-SLEEP DISTURBANCE - SF 8A
Sleep Quality | Third week: mid-treatment (after second session)
  PROMIS-SLEEP DISTURBANCE - SF 8A
Sleep Quality | Fifth week: post-treatment (after fourth session)
  PROMIS-SLEEP DISTURBANCE - SF 8A
Sleep Quality | 4 months: 3 month follow-up
  PROMIS-SLEEP DISTURBANCE - SF 8A
Illness Perception | Assessed via telephone within a 1-week period at baseline (prior to randomization)
  Illness Perception Questionnaire
Illness Perception | Third week: mid-treatment (after second session)
  Illness Perception Questionnaire
Illness Perception | Fifth week: post-treatment (after fourth session)
  Illness Perception Questionnaire
Illness Perception | 4 months: 3 month follow-up
  Illness Perception Questionnaire

OTHER OUTCOMES:
Medication use for Fatigue | Assessed via telephone within a 1-week period at baseline (prior to randomization)
  CO-VARIATE - Medication self-report
Medication use for Fatigue | Third week: mid-treatment (after second session)
  CO-VARIATE - Medication self-report
Medication use for Fatigue | Fifth week: post-treatment (after fourth session)
  CO-VARIATE - Medication self-report
Medication use for Fatigue | 4 months: 3 month follow-up
  CO-VARIATE - Medication self-report

CONTACTS AND LOCATIONS:
Overall Officials: M. Elena Mendoza, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States